CLINICAL TRIAL: NCT00210743
Title: An Open-Label, Clinical Evaluation of the Initiation of Every 2 Week Epoetin Alfa (PROCRIT)in the Treatment of Subjects With the Anemia of Chronic Kidney Disease (CKD)
Brief Title: Alternate Dosing - Initiation of Every 2 Week Epoetin Alfa (PROCRIT) in the Treatment of Anemia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004600
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Kidney Diseases
Keywords: Anemia; chronic kidney disease; erythropoetin, Epoetin alfa; erythropoetin recombinant; pre-dialysis
MeSH Terms: conditions — Anemia; Kidney Diseases; Renal Insufficiency, Chronic | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the hemoglobin response rate in subjects with anemia, associated with chronic kidney failure, after receiving epoetin alfa (PROCRITÂ®) every 2 weeks

DETAILED DESCRIPTION:
This is a prospective study in non-dialysis subjects with anemia associated with chronic kidney disease. Subjects will be enrolled from multiple centers in the United States. The primary objective of the study is to evaluate hemoglobin response rate. The secondary objectives include evaluating the time to when hemoglobin responds, indicated by the results of the hemoglobin blood levels, the change in hemoglobin over time, the transfusion requirements and change in quality of life measurements. These measurements asks for the subjects views about how one feels, activity and energy level, etc. The subjects are administered study drug every 2 weeks through Study Week 27 unless dosing is held or the subject withdraws from the study. Each injection of study drug should not exceed 1 ml in volume.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic kidney disease and a glomerular filtration rate within 10-60 ml/min/1.73m2 with no expected need for dialysis during the study
* subjects with a hemoglobin less than 11 g/dL
* subjects who have not received erythropoietic agents within 6 weeks before study entry
* female subjects, with a reproductive potential, must have a negative urine pregnancy test within 7 days of the first dose of study drug.

Exclusion Criteria:

* Subjects with poorly controlled high blood pressure (hypertension) - systolic > 150 mm Hg or diastolic > 100 mm Hg
* known hypersensitivity to human albumin and/or mammalian cell-derived products
* subjects receiving dialysis
* subjects with a ferritin level < 50 ng/mL, Transferrin Saturation < 20%
* subjects receiving chemotherapy for cancer within 1 month prior to study start or expected during study participation
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2004-05; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the number of subjects who achieve a hemoglobin response after receiving PROCRIT every 2 weeks. Hemoglobin response is defined as achieving a target hemoglobin range of 11-12 g/dL for at least 2 consecutive weeks by Week 28.

SECONDARY OUTCOMES:
The secondary endpoints include: the time to a hemoglobin response, the number of subjects achieving a 1 g/dL rise in hemoglobin, change in quality of life measurements, and the total study drug dose up to the time of response.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Benz R, Schmidt R, Kelly K, Wolfson M. Epoetin alfa once every 2 weeks is effective for initiation of treatment of anemia of chronic kidney disease. Clin J Am Soc Nephrol. 2007 Mar;2(2):215-21. doi: 10.2215/CJN.02590706. Epub 2007 Jan 10. PMID 17699416
- See also: An Open-Label, Clinical Evaluation of the Initiation of Every 2 Week PROCRIT (epoetin alfa) in the Treatment of Subjects with the Anemia of Chronic Kidney Disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=604&filename=CR004600_CSR.pdf